CLINICAL TRIAL: NCT04969341
Title: Improving Lung Cancer Screening Barriers for Vulnerable Populations
Brief Title: Improving Lung Cancer Screening Adherence by Overcoming Barriers for Vulnerable Populations
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 21G.139; JT 16804 (Other: JeffTrial Number)
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening (survey, medical record review): Patients complete survey over 20 minutes consisting of validated and piloted items related to cost and convenience barriers in lung cancer screening, personal financial and lung cancer risk perception questions, and the Telehealth Satisfaction and Usefulness questionnaire. Patients also have their medical records reviewed retrospectively.
  Interventions: Other: Survey Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Survey Administration — Complete survey
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study investigates multi-level barriers to lung cancer screening uptake and adherence to lung cancer screening. Identifying cost- and convenience-related barriers to lung cancer screening may help researchers develop targeted strategies to facilitate screening adherence specifically among vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the Jefferson LCSP and eligible for lung cancer screening by our standard criteria (United States Preventive Services Task Force, Center for Medicaid and Medicare Services, and/or National Comprehensive Cancer Network group II guidelines) will be eligible for inclusion in the study
* Additionally, individuals must provide a signed and dated informed consent form to participate in the survey portion of this study

Exclusion Criteria:

* Non-English-speaking individuals
* Individuals who lack consent capacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the Jefferson Lung Cancer Screening Program (LCSP) and eligible for lung cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 947 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Associations between health insurance availability and financial burdens as factors in lung cancer screening adherence | Up to study completion; 15 months
  Individual-level insurance status will be analyzed for association with lung cancer screening adherence. Descriptive analyses of neighborhood factors will be conducted to characterize residential computed tomography (CT)s. Multilevel logistic regression models examining the relationship between screening adherence and each neighborhood factor (i.e., one per model for each CT) and will be adjusted for important individual-level covariates, such as patient age, sex, and smoking status. To address the dependence of the neighborhood factors on race in predicting screening adherence, the modeling results will be focused on interaction terms to examine interactions between race and neighborhood factors.
Individual-level cost-related factors associated with screening adherence | Up to study completion; 15 months
  Will use generalized linear mixed effects logistic regression to model the longitudinal adherence to lung cancer screening as a function of cost-related variables, race, and their interactions. The model will be used to estimate odds ratios representing how adherence associated with financial variables depends on race at each follow-up CT scan.
Convenience-related factors that impact lung cancer screening adherence | Up to study completion; 15 months
  Will assess convenience-related factors that may affect lung cancer screening uptake and adherence. Survey items will address technology and internet accessibility; preferred methods for patient communication; effectiveness of patient navigation; and identification of logistical barriers along each step of the screening workflow including referral, eligibility assessment, scheduling, shared decision-making (SDM) visit, low dose CT (LDCT), results review, and follow-up instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No